CLINICAL TRIAL: NCT03122912
Title: Explore Effects of Dietary Fish Oil in Human Skin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment and interactions/interventions paused due to COVID-19. Not expected to resume in the future. This is not a suspension of IRB approval
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gary Fisher, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00113555 / Derm 683
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Aging Problems
Keywords: fish oil
MeSH Terms: interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish Oil (Experimental): Capsules contain omega-3 fatty acids (fish oil). Dosage of 3180 mg of omega-3 fatty acids will be taken orally daily up to 16 weeks.
  Interventions: Dietary Supplement: Fish Oil
- Soybean Oil (Active Comparator): Dosage will be 3000 mg of soybean oil taken orally daily for up to 16 weeks.
  Interventions: Dietary Supplement: Soybean Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Capsules contain omega-3 fatty acids (fish oil). Dosage of 3180 mg of omega-3 fatty acids will be taken orally daily up to 16 weeks.
  Arms: Fish Oil
Dietary Supplement: Soybean Oil — Dosage will be 3000 mg of soybean oil taken orally daily for up to 16 weeks.
  Arms: Soybean Oil

SUMMARY:
The purpose of this study is to explore the potential differences in the skin of people who take fish oil versus soybean oil pills.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age.
* Good general health.
* No disease states or physical conditions, which would impair evaluation of the biopsy sites.
* Signed, written and witnessed, Informed Consent Form
* BMI is between 18 to 36 kg/m2

Exclusion Criteria:

* Pregnant or lactating women or women contemplating pregnancy for the duration of the protocol. A pregnant test will not be given to women who are capable to pregnant.
* Lovaza™ (prescription fish oil) and not willing to go off Lovaza for 3 weeks prior to enrollment to end of study.
* Frequent NSAID use (not including low dose aspirin) and not willing to go off NSAIDS for 3 weeks prior to enrollment and to end of study.
* Steroids (except inhaled steroids for asthma) and not willing to go off steroids for 3 weeks prior to enrollment to end of study.
* Other medications that may affect the biomarkers of interest.
* Any supplement use (i.e. fish oils, flax seed oils and other oils) that can affect the biomarkers of interest.
* Diet with frequent (1-2 days per week) oily fish (mackerel, salmon, sardines, cold water fish, et al).
* History of photosensitive conditions (connective tissue diseases, polymorphous light eruption, porphyrias etc).
* Received an experimental drug or used experimental device in the 30 days prior to admission to the study.
* History of keloids or any other condition that would complicate wound healing.
* Allergic to soybean, soybean oil, peanuts or seafood.
* History of allergic reactions to local anesthetics.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in barrier function improvement from Baseline to Week 16. | 16 weeks
  Barrier function will be measured at baseline and 16 weeks. Differences in barrier function between the two visits will be assessed.
Number of subjects with barrier function improvement from Baseline to Week 16. | 16 weeks
  Barrier function will be measured at baseline and 16 weeks. The number of subjects with dichotomized improvement in barrier function between the two visits will be compared.

SECONDARY OUTCOMES:
Change in Omega-3 Fatty Acid Levels in blood from Baseline to Week 16. | 16 weeks
  Omega-3 fatty acids in blood will be measured at baseline and 16 weeks. Differences in levels between the two visits will be assessed.
Number of subjects with increased Omega-3 Fatty Acid Levels in Blood from Baseline to Week 16. | 16 weeks
  Omega-3 fatty acids in blood will be measured at baseline and 16 weeks. The number of subjects with dichotomized improvement in levels between the two visits will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fisher, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black HS, Rhodes LE. Potential Benefits of Omega-3 Fatty Acids in Non-Melanoma Skin Cancer. J Clin Med. 2016 Feb 4;5(2):23. doi: 10.3390/jcm5020023. PMID 26861407
- [Background] Millsop JW, Bhatia BK, Debbaneh M, Koo J, Liao W. Diet and psoriasis, part III: role of nutritional supplements. J Am Acad Dermatol. 2014 Sep;71(3):561-9. doi: 10.1016/j.jaad.2014.03.016. Epub 2014 Apr 26. PMID 24780177
- [Background] Pilkington SM, Rhodes LE, Al-Aasswad NM, Massey KA, Nicolaou A. Impact of EPA ingestion on COX- and LOX-mediated eicosanoid synthesis in skin with and without a pro-inflammatory UVR challenge--report of a randomised controlled study in humans. Mol Nutr Food Res. 2014 Mar;58(3):580-90. doi: 10.1002/mnfr.201300405. Epub 2013 Dec 5. PMID 24311515
- [Background] Rhodes LE, Shahbakhti H, Azurdia RM, Moison RM, Steenwinkel MJ, Homburg MI, Dean MP, McArdle F, Beijersbergen van Henegouwen GM, Epe B, Vink AA. Effect of eicosapentaenoic acid, an omega-3 polyunsaturated fatty acid, on UVR-related cancer risk in humans. An assessment of early genotoxic markers. Carcinogenesis. 2003 May;24(5):919-25. doi: 10.1093/carcin/bgg038. PMID 12771037
- [Background] Rhodes LE, Durham BH, Fraser WD, Friedmann PS. Dietary fish oil reduces basal and ultraviolet B-generated PGE2 levels in skin and increases the threshold to provocation of polymorphic light eruption. J Invest Dermatol. 1995 Oct;105(4):532-5. doi: 10.1111/1523-1747.ep12323389. PMID 7561154
- [Background] Rhodes LE, O'Farrell S, Jackson MJ, Friedmann PS. Dietary fish-oil supplementation in humans reduces UVB-erythemal sensitivity but increases epidermal lipid peroxidation. J Invest Dermatol. 1994 Aug;103(2):151-4. doi: 10.1111/1523-1747.ep12392604. PMID 8040603
- [Background] Vargas ML, Almario RU, Buchan W, Kim K, Karakas SE. Metabolic and endocrine effects of long-chain versus essential omega-3 polyunsaturated fatty acids in polycystic ovary syndrome. Metabolism. 2011 Dec;60(12):1711-8. doi: 10.1016/j.metabol.2011.04.007. Epub 2011 Jun 2. PMID 21640360
- [Background] Shinto L, Marracci G, Mohr DC, Bumgarner L, Murchison C, Senders A, Bourdette D. Omega-3 Fatty Acids for Depression in Multiple Sclerosis: A Randomized Pilot Study. PLoS One. 2016 Jan 22;11(1):e0147195. doi: 10.1371/journal.pone.0147195. eCollection 2016. PMID 26799942
- [Background] Tecklenburg-Lund S, Mickleborough TD, Turner LA, Fly AD, Stager JM, Montgomery GS. Randomized controlled trial of fish oil and montelukast and their combination on airway inflammation and hyperpnea-induced bronchoconstriction. PLoS One. 2010 Oct 18;5(10):e13487. doi: 10.1371/journal.pone.0013487. PMID 20976161
- [Background] Mozurkewich EL, Clinton CM, Chilimigras JL, Hamilton SE, Allbaugh LJ, Berman DR, Marcus SM, Romero VC, Treadwell MC, Keeton KL, Vahratian AM, Schrader RM, Ren J, Djuric Z. The Mothers, Omega-3, and Mental Health Study: a double-blind, randomized controlled trial. Am J Obstet Gynecol. 2013 Apr;208(4):313.e1-9. doi: 10.1016/j.ajog.2013.01.038. PMID 23531328
- [Background] Flock MR, Skulas-Ray AC, Harris WS, Gaugler TL, Fleming JA, Kris-Etherton PM. Effects of supplemental long-chain omega-3 fatty acids and erythrocyte membrane fatty acid content on circulating inflammatory markers in a randomized controlled trial of healthy adults. Prostaglandins Leukot Essent Fatty Acids. 2014 Oct;91(4):161-8. doi: 10.1016/j.plefa.2014.07.006. Epub 2014 Jul 17. PMID 25091379